CLINICAL TRIAL: NCT04807296
Title: Thulium Fiber Laser Compared to Holmium:YAG Laser With Moses Technology for Enucleation of the Prostate: A Prospective Study
Brief Title: Thulium Fiber Laser Enucleation of the Prostate (TFLEP) vs HoLEP With Moses Technology (m-HoLEP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-02-2021-9505
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Lasers, Solid-State; Lower Urinary Tract Symptoms; Hyperplasia; Urological Manifestations; Prostatic Disease
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Hyperplasia; Urological Manifestations; Prostatic Diseases

STUDY DESIGN:
Intervention Model Description: Each arm will consist of 50 patients: one undergoing Thulium Fiber Laser Enucleation of the Prostate (TFLEP) and the other undergoing Holmium:YAG Laser Enucleation of the Prostate with Moses Technology (m-HoLEP).Two surgeons will be involved in this study. One surgeon with experience with TFLEP will perform all 50 TFLEP procedures and one surgeon with experience with m-HoLEP will perform all 50 m-HoLEP procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TFLEP (Active Comparator): Thulium fiber laser (TFL) is a novel laser technology that delivers a pulsed laser at a more optimal wavelength and a shallower depth of tissue penetration leading to better hemostatic properties. Patients will undergo thulium fiber laser enucleation of the prostate (TFLEP) at the Centre Hospitalier de l'Université de Montréal (CHUM) as a treatment for benign prostate hyperplasia. The surgeon performing TFLEP is experienced in TFLEP procedures.
  Interventions: Procedure: TFLEP
- m-HoLEP (Active Comparator): The holmium: yttrium-aluminum-garnet (Ho: YAG) laser is the longest running and most studied laser used to perform this minimally invasive procedure. Holmium laser enucleation of the prostate reduces hospital stay and hemoglobin drop while improving IPSS and quality of life, as well as other positive postoperative outcomes compared to the historical gold standard, transurethral resection of the prostate (TURP). HoLEP has been found to have a better enucleation efficiency rate and may have better hemostatic properties when combined with the modulated pulsed laser energy featured associated with Moses technology (m-HoLEP). Patients will undergo m-HoLEP at the Centre intégré universitaire de santé et de services sociaux (CIUSSS) du Nord-de-l'Île-de-Montréal as a treatment for benign prostate hyperplasia. The surgeon performing m-HoLEP is experienced in m-HoLEP procedures.
  Interventions: Procedure: m-HoLEP

INTERVENTIONS:
Procedure: TFLEP — Thulium fiber laser (TFL) is a novel laser technology that delivers a pulsed laser at a more optimal wavelength and a shallower depth of tissue penetration leading to better hemostatic properties. Patients will undergo thulium fiber laser enucleation of the prostate (TFLEP) at the Centre Hospitalier de l'Université de Montréal (CHUM) as a treatment for benign prostate hyperplasia. The surgeon performing TFLEP is experienced in TFLEP procedures.
  Fifty (50) patients will undergo TFLEP.
  Arms: TFLEP
Procedure: m-HoLEP — The holmium: yttrium-aluminum-garnet (Ho: YAG) laser is the longest running and most studied laser used to perform this minimally invasive procedure. Holmium laser enucleation of the prostate reduces hospital stay and hemoglobin drop while improving IPSS and quality of life, as well as other positive postoperative outcomes compared to the historical gold standard, transurethral resection of the prostate (TURP). HoLEP has been found to have a better enucleation efficiency rate and may have better hemostatic properties when combined with the modulated pulsed laser energy featured associated with Moses technology (m-HoLEP). Patients will undergo m-HoLEP at the Centre intégré universitaire de santé et de services sociaux (CIUSSS) du Nord-de-l'Île-de-Montréal as a treatment for benign prostate hyperplasia. The surgeon performing m-HoLEP is experienced in m-HoLEP procedures.
  Fifty (50) patients will undergo m-HoLEP
  Arms: m-HoLEP

SUMMARY:
Enucleation of the prostate equips technology (usually laser) to effectively treat lower urinary tract symptoms associated with benign prostate hyperplasia (BPH). The holmium: yttrium-aluminum-garnet (Ho: YAG) laser is considered the gold standard laser used to perform enucleation of the prostate. Holmium laser enucleation of the prostate (HoLEP) reduces hospital stay and hemoglobin drop while improving International Prostate Symptom Score (IPSS) and quality of life, as well as other postoperative outcomes. HoLEP has been found to have a better enucleation efficiency rate and may have better hemostatic properties when combined with the modulated pulsed laser energy featured associated with Moses technology (m-HoLEP).

A novel laser technology called thulium fiber laser (TFL) delivers a pulsed laser at a more optimal wavelength and a shallower depth of tissue penetration leading to better hemostatic properties. However, the differences in clinical outcomes between TFL enucleation of the prostate (TFLEP) and m-HoLEP have yet to be described. This prospective study aims to compare the safety profile and clinical outcomes, peri-operatively up to one year post-operatively, between m-HoLEP and TFLEP with BPH and evidence of bladder obstruction.

DETAILED DESCRIPTION:
Enucleation of the prostate equips technology (usually laser) to effectively treat lower urinary tract symptoms associated with benign prostate hyperplasia (BPH). The holmium: yttrium-aluminum-garnet (Ho: YAG) laser is the longest running and most studied laser used to perform this minimally invasive procedure.

Holmium laser enucleation of the prostate (HoLEP) reduces hospital stay and hemoglobin drop while improving IPSS and quality of life, as well as other positive postoperative outcomes. HoLEP has been found to have a better enucleation efficiency rate and may have better hemostatic properties when combined with the modulated pulsed laser energy featured associated with Moses technology (m-HoLEP).

A novel laser technology called thulium fiber laser (TFL) delivers a pulsed laser at a more optimal wavelength and a shallower depth of tissue penetration leading to better hemostatic properties. However, the differences in clinical outcomes between TFL enucleation of the prostate (TFLEP) and m-HoLEP, to our knowledge, have yet to be described.

This prospective study aims to compare the safety profile and clinical outcomes, peri-operatively up to one year post-operatively, between m-HoLEP and TFLEP with BPH and evidence of bladder obstruction. Variables of particular interest include the length of hospital stay and the need for blood transfusion, which are benefits of both techniques compared to transurethral resection of the prostate, the current gold standard of BPH treatment according to American Urological Association (AUA) guidelines. The results of this study will guide urologists in selecting the most appropriate procedure from the growing armamentarium of treatments for BPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic benign prostate hyperplasia : urinary retention, acute renal failure (post-renal), refractory hematuria, repeated urinary tract infections, refractory symptoms.
* Prostates between 50-300 grams,
* IPSS ≥ 8,
* Inadequate response to previous medical treatments,
* Qmax < 15 ml/sec and
* Providing informed consent

Exclusion Criteria:

* History of prostatic surgery,
* History of prostate or bladder cancer,
* Neurogenic bladder,
* Urethral stricture,
* Anticoagulant therapy (aspirin permitted), not ceased during surgery
* Patients unfit for surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
To compare the hospital stay between the thulium fiber laser enucleation of the prostate (TFLEP) and the holmium:YAG laser enucleation of the prostate with Moses technology (m-HoLEP). | 1 day post-operatively
  Length of hospital stay following surgery, measured in hours and minutes.

SECONDARY OUTCOMES:
To compare intraoperative adverse events between cohorts | During surgery
  Incidence of bleeding and blood transfusion, injury or perforation of the bladder or urinary tract
To compare enucleation and morcellation time between cohorts | During surgery
  Enucleation time and morcellation time, measured in minutes.
To compare enucleation rate of instrumentation between cohorts | During surgery
  Enucleation rate, measured in enucleated tissue (mL) / time (minutes)
To compare operative time between cohorts | During surgery
  Operative time, measured in hours
To compare catheterization time between cohorts | Up to 7-days post-operatively
  Time until catheter was removed from participant post-surgery, measured in hours and minutes
To compare drop in International Prostate Symptom Score (I-PSS) between cohorts | Up to 1-year post-operatively
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
To measure increase of Quality of life (QoL) between cohorts | Up to 1-year post-operatively
  IPSS includes one question pertaining to QoL which asks: "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? Scored from 0-6 with 0 being "delighted" and 6 being "terrible". Higher the score, the lower the quality of life.
To compare peak urine flow rates (Qmax) between cohorts | Up to 1-year post-operatively
  Indicates the maximum urine flow rate. In men peak flow rates (Qmax) less than 15 ml/second are considered abnormal. This is measured by uroflowmetry, which measures the flow and force of urine stream during urination.
To compare change in erectile function (IIEF) between cohorts | Up to 1-year post-operatively
  The International Index of Erectile Function (IIEF) is standardised and validated 15-item self-evaluation scale provides pre-post treatment clinic evaluations of erectile function, orgasmic function, sexual desire, satisfaction in sexual intercourse and general satisfaction.
To compare post-void residual urine volume (PVR) between cohorts | Up to 1-year post-operatively
  Amount of urine retained in the bladder after a voluntary void.
To compare the impact of incontinence (ICIQ-short form) between cohorts | Up to 1-year post-operatively
  The International Consultation on Incontinence Modular Questionnaire - Short Form (ICIQ-SF) reflects the impact of urinary incontinence on QoL. Three (3) items are summed up (frequency of urinary incontinence, amount of leakage, overall impact of urinary incontinence) to provide a score between 0 & 21. Higher scores reflect increased urinary incontinence and poorer QoL.
To compare prostate-specific antigen (PSA) levels between cohorts | Up to 1-year post-operatively
  PSA levels
To compare postoperative complications levels between cohorts | Up to 1-year post-operatively
  Incidence of urinary tract infection and stress or urge incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual data. We do plan to present our findings at conferences however all patient information will be anonymized.